CLINICAL TRIAL: NCT03261219
Title: Intrapulmonary Percussive Ventilation vs Chest Physiotherapy Vest in Airway Clearance During Cystic Fibrosis Pulmonary Exacerbation
Brief Title: IPV vs CPT for Airway Clearance During CF Exacerbation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Not renewed with IRB
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB201700115
Record Dates: First submitted 2017-08-22; First posted 2017-08-24 (Actual); Last update posted 2018-10-19 (Actual); Status verified 2018-10

CONDITIONS: Cystic Fibrosis; Airway Clearance Impairment
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Intrapulmonary Percussive ventilation (Experimental)
  Interventions: Device: Intrapulmonary Percussive ventilation
- Chest Physiotherapy vest (Active Comparator)
  Interventions: Device: Chest Physiotherapy Vest (Incourage)

INTERVENTIONS:
Device: Intrapulmonary Percussive ventilation — mode of airway clearance using mouthpiece and alternating air currents applied directly to the airway
  Arms: Intrapulmonary Percussive ventilation
Device: Chest Physiotherapy Vest (Incourage) — mode of airway clearance using external vibratory vest
  Arms: Chest Physiotherapy vest

SUMMARY:
Intrapulmonary Percussive Ventilation (IPV) will show greater improvements in Forced Expiatory Volume in 1 second (FEV1) shorter duration of stay, and greater time to next pulmonary exacerbation in pediatric Cystic Fibrosis patients admitted for pulmonary exacerbation.

FEV1 is a measurement of obstruction in the airway which is seen to be elevated in CF patients with worsening lung disease. FEV1 is used as a primary endpoint in pulmonary trials because it is an acute indicator of worsening or improving lung function.

DETAILED DESCRIPTION:
The study will be a prospective randomized clinical trial. All Cystic Fibrosis (CF) patients five years and above who are being admitted to University of Florida (UF) Shands Children's Hospital with the diagnosis of CF acute pulmonary exacerbations will be approached for study consent on day one of hospitalization.

Each patient will be randomized to receive either IPV (metaneb) or Chest Physiotherapy (CPT) vest (Incourage) therapy. Treatments will be administered by in-house respiratory therapists four times daily according to standard protocol, and the respiratory therapist will document each treatment in the patient's electronic medical record (EPIC). Each patient will also receive mucolytic agents (dornase alpha, hypertonic saline) and antibiotic therapy as per routine inpatient protocol per the attending pulmonologist on service. If the patient's clinical status worsens during their admission the attending pulmonologist will be allowed to change the airway clearance regimen or antibiotic coverage at their discretion.

If a patient is enrolled and has another admission for pulmonary exacerbation after their initial admission, we will attempt to randomize them to the other arm and utilize this data to see if there is a difference in outcome parameters for the same patient if they are randomized to both arms.

The degree of improvement in FEV1 defined as absolute difference between admission FEV1 and discharge FEV1 will be used as primary outcome measure to compare effectiveness between both modalities. This measure is commonly used in the Cystic Fibrosis community of clinicians and researchers as measure of airway obstruction and disease severity. We will perform spirometry at least twice, at admission and discharge, on these patients. The patient's spirometry from their office visit on the same day of admission or first spirometry during their admission will count as the initial spirometry. Last spirometry obtained before discharge will be the discharge spirometry. Additional spirometry may be performed during the patient's admission at the attending provider's clinical discretion. We will also use data from these additional spirometry measurements if they take place.

There will be no additional cost incurred by using the IPV device as opposed to standard of care (CPT vest).There is also no increased effort performing IPV treatments from the respiratory therapist performing the treatment or from the patient.

Length of hospital stay in days will be used as a secondary outcome.

Another secondary outcome measure will be the length of time between discharge and subsequent admissions for CF pulmonary exacerbation. We will follow the subject for an additional 6 months after they are enrolled to ascertain the time to next admission and total number of admissions in that time.

Other information that will be accessed through EPIC records will be number of admissions for CF pulmonary exacerbations, airway clearance regimen, radiological data, laboratory results (respiratory cultures, Respiratory Viral Panels, Acid Fast Bacilli cultures, complete Blood counts), vital signs, weight measurements, Bronchoscopy reports, medications used (Orkambi, Kalydeco, antibiotics), and oxygen requirement. All of this information will be collected in the time period of 1 year before study and throughout study,

We will also administer a 2 question questionnaire at the beginning and end of admission to the hospital in order to evaluate the patient/family opinion of the therapy they received during their participation in the study.

ELIGIBILITY:
Inclusion Criteria:

* CF patient admitted for pulmonary exacerbation

Exclusion Criteria:

* Patients who are not able to perform spirometry, patients with neurological impairment (Cerebral Palsy) or severe behavioral problems that precludes consistent use of IPV, patients with pneumothorax or significant hemoptysis, patients who require supplemental oxygen or ventilatory support, or patients whose parents/guardians are not willing to consent will be excluded.

Ages: 5 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2018-07 (Estimated); Primary Completion 2018-08-31 (Estimated); Study Completion 2018-10-30 (Estimated)

PRIMARY OUTCOMES:
FEV1 change | duration of hospital stay (usually 10-14 days)
  change in FEV1 from baseline at admission

SECONDARY OUTCOMES:
time to next admission | from discharge to 6 months after discharge
  time in days to next hospital admission for CF Pulmonary Exacerbation
Patient Satisfaction with airway clearance modality | 10 minutes after each discharge during study period
  survey of satisfaction with prescribed airway clearance modality
Length of admission | usually 10-14 days
  length of admission in days

IPD SHARING:
Plan to Share IPD: No